CLINICAL TRIAL: NCT01890564
Title: Modes of Ventilation During Laparoscopic Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman - Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB12-00783
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bariatric surgery: Patients undergoing bariatric surgery.
  Interventions: Other: Pressure controlled ventilation; Other: Volume controlled ventilation; Other: PRVC ventilation

INTERVENTIONS:
Other: Pressure controlled ventilation — For pressure controlled ventilation, the peak inflating pressure (PIP) is set for each tidal breath.
Other: Volume controlled ventilation — For volume controlled ventilation, the tidal volume is set.
Other: PRVC ventilation — Pressure-regulated, volume-controlled (PRVC) is an auto-regulated pressure-controlled mode of mechanical ventilation with a user-selected tidal volume target.

SUMMARY:
During minimally invasive surgery, a pneumoperitoneum is created to facilitate surgical visualization. Although effective in facilitating the procedure, there are respiratory consequences of the pneumoperitoneum, which significantly increases intra-abdominal pressure (IAP) up to 20 cmH2O. The increased IAP can decrease functional residual capacity and increase closing capacity resulting in increased resistance, decreased compliance, and increased ventilation-perfusion mismatch. In a randomized, cross-over design, this study will evaluate in sequential order, 3 modes of ventilation during laparoscopic bariatric surgery to determine which is better able to support oxygenation and ventilation while limiting the peak inflating pressure (PIP).

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic bariatric surgery requiring intra-arterial blood pressure monitoring, age 14-20 years.

Exclusion Criteria:

* None

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Bariatric surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in heart rate | Baseline to 30 mins.
  Heart rate will be assessed every 5 mins. during each 30 minute mode of ventilation.

SECONDARY OUTCOMES:
Change in blood pressure | Baseline to 30 mins.
  Blood pressure will be recorded every 5 mins. during each 30 minute mode of ventilation.
Blood gas | 30 mins.
  Blood gas will be obtained at the end of each 30 minute mode of ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States